CLINICAL TRIAL: NCT03849313
Title: Multicentre, Randomized, Double-Blind, 3-Arm, Parallel Study to Compare the Pharmacokinetics, Safety and Tolerability of AVT02 to EU-approved and US-licensed Humira® Administered as a Single Dose (40 mg Subcutaneous Injection) in Healthy Adult Volunteers (ALVOPA D FIRST)
Brief Title: Pharmacokinetics, Safety and Tolerability Study of AVT02 to EU-approved and US-licensed Humira (Adalimumab)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AVT02-GL-101
Record Dates: First submitted 2019-02-04; First posted 2019-02-21 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: 3 arm trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AVT02 100mg/mL (Experimental): Biosimilar Adalimumab AVT02
  Interventions: Drug: Adalimumab
- EU-Humira 100mg/mL (Active Comparator): EU Approved Adalimumab originator Humira
  Interventions: Drug: Adalimumab
- US-Humira 100mg/mL (Active Comparator): US licensed Adalimumab originator Humira
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — AVT02, a proposed similar biological product (biosimilar) of Humira which contains adalimumab . Adalimumab is a recombinant, fully human monoclonal immunoglobulin G1 (IgG1) antibody that binds specifically and with high affinity to the soluble and transmembrane forms of tumor necrosis factor (TNF)-α thereby inhibiting the binding of TNF-α with its receptor, and inhibiting TNF -α's biological function.
  Tumor necrosis factor-α is a naturally occurring cytokine that is key to normal inflammatory and immune responses. Elevated levels of TNF-α are found in the synovial fluid of rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis patients and psoriasis plaques and play an important role in both the pathologic inflammation and joint destruction that are hallmarks of these inflammatory diseases
  Other Names: Humira ATC code L04AB04

SUMMARY:
This study has been designed as a multicentre, randomised, double-blind study of AVT02 in healthy adult subjects. The study will assess the PK, safety and tolerability of AVT02 compared to EU-Humira and US licenced Humira (US-Humira), when administered as a single 40 mg SC dose.

DETAILED DESCRIPTION:
AVT02 is being developed as a biosimilar to Humira. EU-Humira and US-Humira have therefore been selected as the active control groups in this study.

This study is designed as a multi-center, randomised, double-blind, 3-arm parallel study of AVT02 compared to EU-Humira and US-Humira in healthy adult subjects. The study is designed to evaluate the PK, safety and tolerability of AVT02 compared to EU-Humira and US-Humira when administered as a single dose (40 mg) SC injection.

Subjects will be randomly assigned with a ratio of 1:1:1 to receive either AVT02 or EU-Humira or US-Humira on a single occasion on study Day 1. Both the site staff assessing the subjects and the subjects themselves will be blinded to the treatments being administered.

The study consists of a screening period, admission and treatment period, assessment period and end of study visit. Subjects will undertake a screening visit between Day -28 and Day -1 to determine eligibility in the study. Those subjects that meet the eligibility criteria will be admitted to the study site on the evening prior to dosing (Day -1) when continued eligibility will be assessed.

On Day 1 prior to dosing, baseline assessments will be performed. Subjects will then be dosed according to the randomization schedule. Following dosing, PK, safety and tolerability assessments will be performed according to the study schedule (Table 6Table 6). Subjects will remain confined to the study site from Day -1 to Day 3 (48 hours post-dose). Subjects will return to the study site on Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 12, Day 15, Day 22, Day 29, Day 36, Day 43, Day 50 and Day 57.

An end of study visit will occur at study Day 64 for final study assessments

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy adult subjects willing to sign a patient information and consent form (PICF) and able to undergo protocol related procedures.
* Age: 18 to 55 years, inclusive.
* Body Mass Index (BMI): 18.5 to 32.0 kg/m2.
* No history or evidence of a clinically significant disorder, condition, or disease that, in the opinion of the investigator would pose a risk to subject safety.
* Resting supine systolic blood pressure of ≤150 mmHg and diastolic blood pressure of ≤90 mmHg. Other vital signs showing no clinically relevant deviations according to the investigator's judgment.
* 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the investigator.
* Negative urine drug screen and negative alcohol breath test at screening and admission.

Exclusion Criteria

* Subjects will be excluded from the study if one or more of the following criterion are applicable:
* Evidence of clinically relevant pathology
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agent(s) used in study.
* Known history of previous exposure to adalimumab or other anti TNF-alpha molecules.
* Subjects with a recent (within 6 months of dosing) infection requiring hospitalisation or intravenous antibiotic use.
* Subjects with a recent (within 4 weeks of dosing) infection requiring oral or systemic antibiotics.
* Subject with a history of recurrent or chronic infections.
* Subject has a positive test for tuberculosis (TB) during screening or a known history of active or latent TB, except documented and complete adequate treatment of TB.
* Having received live vaccines during the 4 weeks before screening or have the intention to receive vaccination during the study.
* Participation in a drug study within 60 days or 5 half-lives of the previous drug (if known), whichever is longer, prior to drug administration Note: Only the few inclusion/exclusion criteria are mentioned here. Subjects will be screened and randomized as per the full list of inclusion and exclusion criteria in the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 390 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve AUC0-t | From baseline to day 64
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC 0-t) of AVT02, US-Humira EU Humira
Maximum serum concentration | From baseline to day 64
  Venous blood samples will be collected for measurement of serum concentration of AVT02, EU Humira, US-Humira
Area under the plasma concentration-time curve AUC0-inf | From baseline to day 64
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUC 0-inf) of AVT02, US-Humira EU Humira

SECONDARY OUTCOMES:
Pain, Tenderness, Erythema and Swelling | From baseline to over a 64 day period
  The injection sites will be monitored for pain, tenderness, erythema and swelling. Each injection site reaction will be categorised using the Injection Site Intensity Grading Scheme. All four outcome measures mentioned in the title will be measured from this one scheme.
Anti Drug Antibodies (ADRs) | Baseline to over a 64 day period
  Formation of Anti Drug Antibody will be measured through a validated assay.
Adverse Events | From screening to day 64.
  Adverse events will be coded using MedDRA and grouped by system organ class and preferred term and summarised, by treatment group at the time of onset of the AE. The summary tables will present the number and percentage of total subjects and number of events, by system organ class and by preferred term. Injection related reactions will be listed and summarised by reaction using frequency counts and percentage, by treatment group.
Neutralizing Antibodies (NAbs) | From screening to day 64.
  Formation of neutralizing antibodies measured through a validated system

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schwabe, Principal Investigator — Auckland Clinical Studies Limited
Locations (3):
- Scientia Clinical Research, Sydney, New South Wales, Australia
- New Zealand (2):
  - Christchurch Clinical Studies Trust Limited, Christchurch, Chistchurch
  - Auckland Clinical Studies, Auckland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wynne C, Schwabe C, Lemech C, Stroissnig H, Dias R, Sobierska J, Guenzi E, Otto H, Sattar A, Kay R, Haliduola HN, Berti F. A randomized, adaptive design, double-blind, 3-arm, parallel study assessing the pharmacokinetics and safety of AVT02, a high-concentration (100 mg/mL) Adalimumab biosimilar, in healthy adult subjects (ALVOPAD FIRST). Expert Opin Investig Drugs. 2022 Sep;31(9):965-976. doi: 10.1080/13543784.2022.2035359. Epub 2022 Feb 10. PMID 35107050